CLINICAL TRIAL: NCT04694963
Title: A Integration of Respiratory Medicine and Prevention Multi-center Study to Determine the Prevalence and Influence of Pertussis on Subacute Cough in Shenzhen by National Respiratory Diseases Clinical Medicine Research Center
Brief Title: A Multi-center Study to Determine the Prevalence and Influence of Pertussis on Subacute Cough in Shenzhen
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: WLW-SC-Pertussis
Record Dates: First submitted 2020-12-24; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Pertussis; Chronic Cough
MeSH Terms: conditions — Whooping Cough; Chronic Cough | interventions — Blood Specimen Collection; Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Throat swab, Peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subaute Cough: N=500
  Interventions: Procedure: Blood sample; Procedure: Data collection; Procedure: Throat swab

INTERVENTIONS:
Procedure: Blood sample — 2 ml venous blood was collected and separated into serum.
Procedure: Data collection — 1. Whether the patient has been vaccinated with DPT vaccine and record the time of vaccination;
  2. Medication situation of patients in the past year, including rescue drugs, antitussive and expectorant drugs, inhaled corticosteroids and antibiotics;
Procedure: Throat swab — Before the collection of oropharyngeal swabs, instruct the patient to wash the mouth or gargle, fix the patient's head, open the mouth and expose the throat. If necessary, use a tongue depressor to gently press the tongue.
  Use the swab to wipe the secretion on both sides of the palatal arch, pharynx and tonsil with a sensitive and gentle action, and quickly withdraw the swab to avoid contacting other parts of the mouth.
  Put the swab in the sterile test tube, plug the opening with cotton ball, and send it for inspection and registration in time.

SUMMARY:
A prospective, multi-center, observational clinical trail. Aim to evaluate the real incidence of COPD pertussis and the impact of pertussis on subaute cough.

DETAILED DESCRIPTION:
1. Investigate the incidence and epidemiological characteristics of pertussis infection in subaute cough population.
2. To explore the relationship between pertussis infection and subaute cough.

ELIGIBILITY:
Inclusion Criteria:

* The cough lasts 3 to 8 weeks and there is no obvious evidence of lung disease on chest X-ray.

Exclusion Criteria:

* 1. Major diseases except subaute cough; 2. Significant abnormality in laboratory examination; 3. Clinical diagnosis of lung cancer, bronchiectasis, pneumoconiosis or other simple restrictive ventilation dysfunction; 4. Patients with a history of asthma, allergic rhinitis, or a blood eosinophil count of 2600/mm3 (0.6x10^9/L) within 4 weeks; 5. Currently suffering from active tuberculosis; 6. Patients with life-threatening pulmonary embolism, or al-antitrypsin deficiency, or cystic fibrosis; 7. Patients who have undergone lung resection.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic cough in Shenzhen
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the prevalence of pertussis among subacute cough | Day 0 of each subject at the time of enrollment.
  According to the positive rate of bordetella pertussis nucleic acid, evaluate the prevalence of pertussis in subaute cough.
Evaluation of the correlation between pertussis and subacute cough | Day 0 of each subject at the time of enrollment.
  Evaluate the correlation between pertussis infection and subacute cough by pertussis positive rate and clinical parameters.

SECONDARY OUTCOMES:
Evaluation of the seroprevalence of bordetella pertussis in subacute cough | Day 0 of each subject at the time of enrollment.
  According to anti-pertussis (anti-PT) antibody levels, assess the overall seroprevalence of bordetella pertussis in subacute cough.
Evaluation of the cut-off value for serological diagnosis of pertussis. | Day 0 of each subject at the time of enrollment.
  By comparing the nucleic acid and antibody levels of Bordetella pertussis to evaluate the antibody cut-off value for serological diagnosis of pertussis.
Evaluation of the subtype of bordetella pertussis. | Day 0 of each subject at the time of enrollment.
  According to the level and pattern of different anti-pertussis antibodies (anti-PT, anti-FHA, anti-PRN, anti-FIM2, anti-FIM3), assess the subtype of Bordetella pertussis.

CONTACTS AND LOCATIONS:
Overall Officials: Lingwei Wang, Study Director — Shenzhen People's Hospital
Locations (26):
- China (26):
  - Fuyong people's Hospital of Baoan District, Shenzhen, Shenzhen
  - General Hospital of Shenzhen University, Shenzhen
  - Longhua Branch of Shenzhen People's Hospital, Shenzhen
  - Nanshan District People's Hospital, Shenzhen
  - Peking university shenzhen hospital, Shenzhen
  - Shenzhen Bao'an District Central Hospital, Shenzhen
  - Shenzhen Bao'an District People's Hospital, Shenzhen
  - Shenzhen Hospital of Beijing University of traditional Chinese Medicine, Shenzhen
  - Shenzhen Hospital of Southern Medical University, Shenzhen
  - Shenzhen Hospital of the University of Hong Kong, Shenzhen
  - Shenzhen Longgang District Central Hospital, Shenzhen
  - Shenzhen Longgang District People's Hospital, Shenzhen
  - Shenzhen Longgang District Second People's Hospital, Shenzhen
  - Shenzhen Longgang District Third People's Hospital, Shenzhen
  - Shenzhen Longhua District Central Hospital, Shenzhen
  - Shenzhen Longhua District People's Hospital, Shenzhen
  - Shenzhen Luohu District People's Hospital, Shenzhen
  - Shenzhen People's Hospital, Shenzhen
  - Shenzhen Pingshan District Hospital of traditional Chinese Medicine, Shenzhen
  - Shenzhen Pingshan District People's Hospital, Shenzhen
  - Shenzhen Qianhai Shekou Free Trade Zone Hospital, Shenzhen
  - Shenzhen Second People's Hospital, Shenzhen
  - Shenzhen TCM Hospital, Shenzhen
  - Shenzhen Yantian District People's Hospital, Shenzhen
  - South University of science and Technology Hospital, Shenzhen
  - The eighth Affiliated Hospital of Sun Yat sen University, Shenzhen

IPD SHARING:
Plan to Share IPD: No